CLINICAL TRIAL: NCT03700983
Title: A Pharmacokinetic Study of PEITC in Nutri-Jelly in Healthy Head and Neck Cancer Survivors
Brief Title: A Pharmacokinetic Study of Nutri-PEITC Jelly in Head and Neck Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dental Innovation Foundation Under Royal Patronage (Other)
Collaborators: Maha Vajiralongkorn Thanyaburi Hospital (Unknown); Mahidol University (Other); Srinakharinwirot University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AOF2.2
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Head and neck cancer survivors - patients who had been diagnosed with cancer of lip, oral cavity, oropharynx and nasopharynx, received treatment and the oncologists had defined them as "complete remission", and having normal physical exam and blood biochemistry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutri-PEITC jelly (Experimental): a single serving of 200 g Nutri-PEITC jelly
  Interventions: Dietary Supplement: Nutri-PEITC jelly

INTERVENTIONS:
Dietary Supplement: Nutri-PEITC jelly — an edible, easily to swallow nutritious gel containing a bioactive compound PEITC

SUMMARY:
This research aims to evaluate the absorption and elimination profile of a bioactive compound PEITC in the matrix of Nutri-jelly - a novel edible nutritious gel. Thus, the investigators conducted a pharmacokinetic study in 12 head and neck cancer survivors. After consumed a serving of Nutri-jelly containing 20 mg PEITC, plasma levels of PEITC at 0, 1, 2, 3, 4, 6, 8, 12 and 24 hours were specifically measured by ammonia derivatization and analyzed by liquid chromatography-mass spectrometry (LC-MS/MS). Non-compartmental pharmacokinetic analysis was performed.

DETAILED DESCRIPTION:
β-phenylethyl isothiocyanate (PEITC) is a phytochemical found in cruciferous vegetables with anti-cancer properties in vitro and in vivo. However, its pharmacokinetic profile in cancer survivors were unknown. A pharmacokinetic study was conducted in head and neck cancer survivors to evaluate the absorption and elimination profile of PEITC in the matrix of Nutri-jelly - a novel edible nutritious gel. Twelve head and neck cancer survivors consumed a serving of Nutri-jelly containing 20 mg PEITC. Plasma levels of PEITC at 0, 1, 2, 3, 4, 6, 8, 12 and 24 hours were specifically measured by ammonia derivatization and analyzed by LC-MS/MS. Non-compartmental pharmacokinetic analysis was performed. Pharmacokinetic parameters including Cmax, Tmax, half-life, clearance were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age 20 or above
* Diagnosed with Head and neck cancer
* Completed radiation or chemotherapy since at least 4 weeks ago
* normal physical exam
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2
* Life expectancy > 3 months
* Normal kidney function evidenced by serum creatinine, blood urea nitrogen (BUN), no kidney stone, no history of renal dialysis
* Normal liver function evidenced by serum bilirubin, aspartate transaminase (AST), alanine amino transferase (ALT)
* not pregnant or breastfeeding
* no psychiatric symptoms
* normal vital sign and normal blood chemistry including complete blood count CBC)
* provide voluntary inform consent

Exclusion Criteria:

* unable to communicate
* reject to take Nutri-jelly
* unable to refrain from vegetable intake for 3 days prior to the test
* take paracetamol during 2 days prior to the test
* body weight less than 35 kg or higher than 65 kg
* oral infection such as Candidiasis interfering with normal oral intake

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-08-06 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of PEITC | Day 0 - Day 1
  Plasma concentration of PEITC during 24 hours after intake of Nutri-jelly will be measured and the highest concentration will be identified.
Time to reach maximum concentration (Tmax) | Day 0 - Day 1
  The duration to reach maximum plasma concentration of PEITC will be calculated.

SECONDARY OUTCOMES:
Area under the curve of plasma concentration of PEITC and time | Day 0 - Day 1
  Graph between plasma concentration and time will be plotted. The area under the curve will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Dunyaporn Trachootham, DDS, PhD, Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No